CLINICAL TRIAL: NCT05846906
Title: Oral Sildenafil Citrate: a Potential Approach for Improvement of Endometrial Thickness and Treatment of Unexplained Infertility in Women
Brief Title: Effect of Oral Sildenafil Citrate on Improvement of Endometrial Thickness
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-21015
Record Dates: First submitted 2023-04-15; First posted 2023-05-06 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Sildenafil Citrate; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil and clomiphene citrate (Experimental): Oral Clomiphene citrate (Tecnovula®) 50 mg was taken twice daily by the experimental group from day 2 through day 7 of the cycle, and oral sildenafil (Respatio® 20mg for 5 days) was taken from the last day of menstruation until reaching ovulation.
  Interventions: Drug: Sildenafil Citrate; Drug: Clomiphene Citrate 50mg
- clomiphene citrate alone (Other): Oral Clomiphene citrate (Tecnovula®) 50 mg was taken twice daily by the control group from day 2 through day 7 of the cycle in addition to a placebo tablet.
  Interventions: Drug: Clomiphene Citrate 50mg

INTERVENTIONS:
Drug: Sildenafil Citrate — oral sildenafil (Respatio® 20mg )
  Other Names: respatio
  Arms: Sildenafil and clomiphene citrate
Drug: Clomiphene Citrate 50mg — used for ovionulation induct
  Other Names: technovula

SUMMARY:
One hundred thirty women with unexplained infertility participated in a prospective clinical study. Patients were assigned at random to one of two groups. The first group (n=65) served as the study group and was given clomiphene citrate 50 mg (Tecnovula®, Techno Pharmaceuticals, Egypt) and sildenafil (Respatio®, Pharma right group, Egypt) 20 mg tablets. The second group (n=65) served as a control and received a placebo tablet in addition to the standard treatment of clomiphene citrate 50 mg (Tecnovula®). A transvaginal ultrasound was performed on all of the patients to assess ovulation.

DETAILED DESCRIPTION:
One hundred thirty women with unexplained infertility participated in a prospective clinical study. Patients were assigned at random to one of two groups. The first group (n=65) served as the study group and was given clomiphene citrate 50 mg (Tecnovula®, Techno Pharmaceuticals, Egypt) orally twice daily from the second day of their cycle through the seventh day and sildenafil (Respatio®, Pharma right group, Egypt) 20 mg tablets from the end of menstruation through ovulation. The second group (n=65) served as a control and received a placebo tablet in addition to the standard treatment of clomiphene citrate 50 mg (Tecnovula®). A transvaginal ultrasound was performed on all of the patients to assess ovulation, follicle count, and pregnancy. Consequences, including miscarriage, ectopic pregnancy, and multiple pregnancies, were monitored.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18 to 40
* patent tubes
* unexplained infertility
* regular menstrual cycle
* husband with normal sperm parameters

Exclusion Criteria:

* hypotension
* cardiovascular, renal and hepatic diseases
* uncontrolled diabetes mellitus
* anovulatory infertility
* abnormal thyroid functions
* ovarian cysts
* patients taking nitrates
* pelvic adhesions
* abnormal hormonal profile.
* hyperprolactinemia
* multiple uterine fibroids
* adenomyosis and endometriosis suspicion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | at the end of the cycle (28 days)
  Serum pregnancy test (positive/negative)

SECONDARY OUTCOMES:
endometrial thickness | 1 month
  measured by trans-vaginal ultrasound
ovulation rate | 1 month
  using trans-vaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Study Director — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No